CLINICAL TRIAL: NCT04308824
Title: Efficacy of Cyanoacrylate in the Prevention of Delayed Bleeding After Endoscopic Mucosal Resection of Large Colorectal Polyps.
Brief Title: Cyanoacrylate to Stop Bleeding After EMR for Large Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 683503
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clipping (Active Comparator): Prophylactic endoscopic clip will be placed after polypectomy
  Interventions: Other: clipping
- Cyanoacrilate (Experimental): A solution of Cyanoacrilate will be nebulized after the placement of prophylactic clip
  Interventions: Other: nebulization of glue

INTERVENTIONS:
Other: clipping — a single clip will be placed in every case of polypectomy for large colorectal polyps
  Arms: Clipping
Other: nebulization of glue — After clipping, a cyanoacrilate glue will be nebulized using a spray catheter
  Arms: Cyanoacrilate

SUMMARY:
Endoscopic resection of large non-pedunculated adenomas is most often performed using the 'lift-and-cut' endoscopic mucosal resection (EMR) technique. This endoscopic technique has a relatively low technical complexity and short-duration and is commonly considered a safe and reliable surgical option, nevertheless several adverse events can occur during or after this procedure.

One of the most frequent late complication is the post-procedural bleeding occurring up to 30 days post-polypectomy, which often requires emergency hospitalization and re-intervention.

Endoscopic hemostasis of active post procedure bleeding can be achieved using prophylactic clips.

Recently, the use on sprayable hemostatic agents have been introduced in the gastrointestinal endoscopical practice.

Cyanoacrylate is a liquid tissue adhesive that has been proved to be of some utility in the endoscopic management of gastrointestinal variceal bleeding.

In this study the investigators aim to compare the rate of postoperative bleeding between two groups of patients with large colorectal polyps. In the first group it will be performed a prophylactic clipping after the polypectomy and in the other group it will be used cyanoacrylate after clipping.

DETAILED DESCRIPTION:
Introduction of endoscopic removal of colorectal polyps in the clinical practice has profoundly contributed to the modified epidemiology of colorectal cancer in western countries by reducing its incidence and mortality through a primary prevention. Endoscopic removal of polyps can be carried out using several techniques depending on their morphology, size, location along the colon and the expertise of the endoscopist.

Endoscopic resection of large non-pedunculated adenomas is most often performed using the 'lift-and-cut' endoscopic mucosal resection (EMR) technique. This endoscopic technique has a relatively low technical complexity and short-duration and is commonly considered a safe and reliable surgical option, nevertheless several adverse events can occur during or after this procedure, even in experienced hands. One of the most frequent late complication is the post-procedural bleeding (PPB) occurring up to 30 days post-polypectomy, which often requires emergency hospitalization and re-intervention (by repeated endoscopy, angiography, or even major surgery). The frequency of PPB after EMR of colonic polyps is reported between 0.4 % and 7 % depending on patients' co-morbidities and medications, location and size of the polyps and endoscopic technique.

Endoscopic hemostasis of active PPB can be achieved using different techniques according to the location and characteristics of the lesion, endoscopist's preference and experience, and device availability. However, the most commonly method used is clipping with or without adrenaline injection.

Recently, the use on sprayable hemostatic agents have been introduced in the gastrointestinal endoscopical practice providing a non-traumatic and technically easy method of hemostasis which can be used also in cases of diffuse, multifocal source of bleeding due to ulcers, tumors or post-EMR or in areas difficult to access, such as the lesser curvature of the stomach, posterior wall of the duodenal bulb.

Cyanoacrylate is a liquid tissue adhesive that has been proved to be of some utility in the endoscopic management of gastrointestinal variceal bleeding.

In this study, we will compare the short and mid-term results of the endoscopic use of N-butyl-2-cyanoacrylate associated with methacryloxysulfolane in the prevention of delayed bleeding after EMR of large colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

* peduncolated or flat polyps > 2cm of the colon
* anticoagulant therapy interrupted 5 days before the procedure

Exclusion Criteria:

* Coagulation disorders
* pregnancy
* malignant appearing polyps

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2022-04-02 (Estimated)

PRIMARY OUTCOMES:
Early bleeding | 24 hours
  Bleeding is defined as early if occurrs within 48h after the procedure
Delayed bleeding | 2-7 days
  Bleeding is defined as delayed if occurrs more than 48 hours after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Martines, MD, Study Chair — DETO
Locations (1):
- Dept of Emergency and Organ transplantation - University of Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No